CLINICAL TRIAL: NCT00692380
Title: A Phase I Dose Intensification Study Using Gated Intensity Modulated Radiation Therapy and Concurrent Chemotherapy for Patients With Inoperable, Non-Small Cell Lung Cancer
Brief Title: Gated Intensity Modulated Radiation Therapy and Concurrent Chemotherapy for Inoperable NSCLC
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: insufficient accrual
Sponsor: Virginia Commonwealth University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCC-10274
Record Dates: First submitted 2008-06-03; First posted 2008-06-06 (Estimated); Last update posted 2016-05-02 (Estimated); Status verified 2016-04

CONDITIONS: Non-small Cell Lung Cancer
Keywords: gated IMRT
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Fractionated Radiation Therapy followed by Carboplatin and Taxol
  Interventions: Radiation: Fractionated radiation therapy followed by chemotherapy

INTERVENTIONS:
Radiation: Fractionated radiation therapy followed by chemotherapy — Increasing doses of radiation therapy

SUMMARY:
Radiation therapy technology that allows increased radiation dose to the tumor while sparing healthy tissue will improve the balance between complications and cure.

DETAILED DESCRIPTION:
The primary objective is to establish the maximum tolerated fractional dose (MTfD) of radiotherapy to a total dose of 78Gy using gated IMRT, delivered in single daily fractions that can be administered concurrently with Taxol® and carboplatin chemotherapy. Secondary objectives include: to evaluate the toxicity of concurrent Taxol® and carboplatin with gated IMRT; identify partial organ tolerance doses for lung and esophagus when treating with involved field thoracic 3D; estimate complete response rate as defined by PET performed 3 months after completion of all therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically-proven, by biopsy or cytology, unresectable lung cancer of the following histologic types: squamous cell carcinoma, adenocarcinoma, large cell carcinoma, non-small cell carcinoma, not otherwise specified.
* Patient with AJCC Stage IIIA-IIIB, if all detectable tumor can be encompassed by radiation therapy fields, including both the primary tumor and the involved regional lymph nodes.
* 18-fluoro-2-deoxyglucose positron emission tomography required for staging and image fusion for treatment planning.
* Atelectasis, if present, must be less than one lung.
* Patients must have granulocytes >1500/µl; platelets >100,000/µl; bilirubin < 1.5 mg/dl; AST(SGOT) < 2 ULN; serum creatinine < 2.0 mg/dl.
* Zubrod Score 0-1.
* FEV1 must be >1.0 L.
* Patients must sign a study-specific informed consent form prior to study entry
* Patients must have measurable disease on the planning CT.
* Patient must have a completed the IMRT plan and the attending physician must have reviewed and approved the dose volume histograms as follows (based on treatment planning to the Phase 4 dose level): total lung V20 < 30%, mean esophageal dose < 34 Gy, the esophageal V55 < 30%, the heart V40 < 50%.
* No prior or concurrent malignancy except non-melanomatous skin cancer unless disease-free for one year or more; no prior lung cancer within last two years.
* No prior RT to thorax.
* No previous chemotherapy or previous biologic response modifiers for current lung cancer or within the past five (5) years.
* No distant metastases or supraclavicular lymph node involvement or significant atelectasis.
* No clinically significant pleural effusions, pericardial effusions or superior vena cava syndrome.

Exclusion Criteria:

* Undifferentiated small cell (oat cell or high grade neuroendocrine) carcinoma, any stage.
* Stage I, II or IV NSCLC.
* Complete tumor resection, recurrent disease, or those patients eligible for definitive surgery.
* Concurrent malignancy except non-melanomatous skin cancer or prior cancer unless disease-free for one year or more.
* Prior radiation therapy to the thorax.
* Previous chemotherapy or previous biologic response modifiers for current lung cancer or within the past five (5) years.
* Distant metastases or supraclavicular lymph node involvement, or atelectasis of an entire lung.
* Patients who have not had the pre-treatment evaluations in Section 4.0 or evaluations performed > 8 weeks prior to study entry.
* Patients with clinically significant pleural effusions, pericardial effusions or superior vena cava syndrome.
* Prior lung cancer within the last two years.
* Patients who have significant atelectasis and in whom the CT definition of the gross tumor volume(GTV) is difficult to determine.
* Pregnant or lactating females. It is not known what effects this treatment may have on the developing fetus.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-06; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 3 years

SECONDARY OUTCOMES:
To identify partial organ tolerance doses for lung and esophagus when treating with involved field thoracic 3D. To estimate complete response rate as defined by PET performed 3 months after completion of all therapy. | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Weiss, M.D., Principal Investigator — Massey Cancer Center
Locations (1):
- Massey Cancer Center, Richmond, Virginia, United States